CLINICAL TRIAL: NCT06073639
Title: The Clinical Effect of Autogenous Dentin Graft in Mandibular Third Molar Surgery
Brief Title: The Efficacy of Autogenous Dentin Graft in Mandibular Wisdom Tooth Extraction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Medicine and Pharmacy at Ho Chi Minh City (Other)
Responsible Party: Principal Investigator, Son Hoang Le, Lecturer, University of Medicine and Pharmacy at Ho Chi Minh City
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: VN01002/IORG00086/FWA0002448
Record Dates: First submitted 2023-09-25; First posted 2023-10-10 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Periodontal Pocket; Swelling Lips & Face; Trismus; Pain, Acute
MeSH Terms: conditions — Periodontal Pocket; Facies; Trismus; Acute Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dentin graft (Experimental)
  Interventions: Procedure: Autogenous dentin graft
- Conventional (No Intervention)

INTERVENTIONS:
Procedure: Autogenous dentin graft — Dentin graft is made from the participant extracted tooth by using Kometa Smart Dentin Grinder
  Arms: Dentin graft

SUMMARY:
The study aimed to investigate clinical effect of autogenous dentin graft on patients following mandibular wisdom tooth extraction. The primary outcomes are pain, swelling, trismus and soft tissue healing index within one week after surgery. The investigators also measured periodontal healing of distal aspect of the adjacent second molar up to 2 year after the surgery.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years old
* Symmetry mandibular third molars
* Symmetry maxillary third molars with no caries or periodontal disease
* Mandibular second molars are available

Exclusion Criteria:

* Systematic health has contraindication for surgery
* Pregnant or breastfeeding women
* Allergy with Lidocaine
* Abnormal signs surrounding mandibular third molars

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2024-02-28 (Estimated)

PRIMARY OUTCOMES:
Rate of self-reported pain | 3 days, 7 days
  Pain is measured by self-reported Likert scale from 0 to 5. Higher score indicated more painful situation. Result is reported by the mean score.
Self-reported swelling | 3 days, 7 days
  Patients reported their perception about swelling levels. There are 6 levels of this scale, score from 0 to 5. Higher score means more swelling.
Trismus | 3 days, 7 days
  Trismus is measured by difference of maximal mouth opening between post-and pre-operative wisdom tooth surgery. Maximal mouth opening is mueasured by distance of mesial incisal edge of maxillary and mandibular central incisor.
Soft tissue healing score | 3 days, 7 days, 30 days
  The soft tissue healing score is evaluated according to Hamzami (2018). It includes 8 sub-items. Each item is recorded as 0 or 1 (score). Then, total score of the first 30 days (3 evaluation time) is used to classify wound healing level (good, acceptable, and bad).
Aveolar height | 7 days, 2 months, 6 months, 2 years
  Aveolar height is measured as the distance from cementoenamel joint on distal surface of second molar to the aveolar ridge. The landmark points are defined on periapical film. The aveolar height is measured at 7 days, 3 months, 6 months and 2 years after the surgery.
Swelling measured by facial dimension | 3 days, 7 days
  Difference of distances of facial landmark points between post-and pre-operative wisdom tooth surgery. Two distances (AB and CD) from 4 landmark points are used for measurement: A - lateral commissure of the eye, B - gonion, C - tragus, and D - lateral commissure of the lips.

CONTACTS AND LOCATIONS:
Overall Officials: Son H Le, Principal Investigator — University of Medicine and Pharmacy at Ho Chi Minh City
Locations (1):
- Son Hoang Le, Ho Chi Minh City, District 5, Vietnam

IPD SHARING:
Plan to Share IPD: Yes